CLINICAL TRIAL: NCT00479336
Title: A Dose-defining Study of OPC-41061 in Treatment of Hepatic Edema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 156-06-005
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Results first posted 2014-03-14 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-01

CONDITIONS: Cirrhosis
Keywords: OPC-41061; Tolvaptan; ascites; Cirrhosis
MeSH Terms: conditions — Fibrosis; Ascites | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator)
  Interventions: Drug: OPC-41061 placebo
- 2 (Experimental)
  Interventions: Drug: OPC-41061 7.5mg
- 3 (Experimental)
  Interventions: Drug: OPC-41061 15mg
- 4 (Experimental)
  Interventions: Drug: OPC-41601 30mg

INTERVENTIONS:
Drug: OPC-41061 7.5mg — 7.5mg, 1 tablet a day
  Arms: 2
Drug: OPC-41061 placebo — placebo, 1 tablet a day
  Arms: 1
Drug: OPC-41061 15mg — 15mg, 1 tablet a day
  Arms: 3
Drug: OPC-41601 30mg — 30mg, 1 tablet a day
  Arms: 4

SUMMARY:
To investigate the dose response for changes from baseline in body weight as a primary endpoint and to investigate improvement in ascites, abdominal circumference, lower-limb edema, and pleural effusion as secondary endpoints in seven-day repeated oral administration of OPC-41061 at 7.5, 15, and 30 mg/day or placebo in cirrhosis patients with ascites despite taking conventional diuretics.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with ascites despite taking either of the following combinations of loop diuretics and an anti-aldosterone agent (spironolactone) for at least 7 days prior to start of the study drug administration.

   Combination 1: Loop diuretics at indicated below in combination with an anti-aldosterone agent at a daily dose of 25 mg or more
   * Furosemide: 40 mg/day or more
   * Other loop diuretic: a daily dosage equivalent to 40 mg or more of furosemide Bumetanide: 1 mg/day or more, Piretanide: 6 mg/day or more, Azosemide: 60 mg/day or more, Torasemide: 8 mg/day or more Combination 2: Anti-aldosterone agent at a daily dose of 50 mg or more in combination with furosemide at a daily dose of 20 mg or more (or one of the other loop diuretics specified in Combination 1 at a daily dosage equivalent to 20 mg or more of furosemide)
2. Patients who have been hospitalized or are able to stay at the study site from the start of the run-in observation period until completion of postdosing observation 2.
3. Subjects capable of giving informed consent to participate in the study of their own free will.

Exclusion Criteria:

1. Subjects with any of the following complications or symptoms: (1) Hepatic encephalopathy (Hepatic coma grade: II or more), (2) Poorly-controlled hepatocellular carcinoma (i.e., hepatocellular carcinoma with vessel infiltration confirmed by imaging in the main trunk or main branch of the portal vein, inferior vena cava, or the main trunk of the hepatic vein), (3)Endoscopic findings within 30 days prior to screening examination requiring new therapy for esophageal and gastric varicose vein during the study period, (4)Repeated haemorrhoidal bleeding due to rectal varicose vein within 30 days prior to screening examination, (5)Diabetes mellitus with poorly controlled blood glucose, (6)Heart failure (NYHA class III or IV), (7)Anuria, (8)Impairment of urination due to urinary tract stricture, urinary calculus, tumor in the urinary tract, or other cause
2. Subjects with a history of any of the following diseases: (1) Cerebrovascular disorder within 30 days prior to the screening examination, (2)Episode of gout within 90 days prior to the screening examination, (3)Hypersensitivity or idiosyncratic reaction to benzazepine derivatives such as mozavaptan hydrochloride or benazepril hydrochloride.
3. Subjects who are obese (body mass index [BMI, body weight (kg)/height (m)2] exceeding 35)
4. Patients with supine systolic blood pressure exceeding 90 mmHg
5. Subjects with any of following abnormal laboratory values: hemoglobin exceeding 8.0 g/dL, total bilirubin exceeding 3.0 mg/dL, serum creatinine exceeding 3.0 mg/dL, serum sodium exceeding 147 mEq/L, serum potassium exceeding 5.5 mEq/L, or uric acid exceeding 8.0 mg/dL
6. Patients who are unable to take oral medication
7. Female subjects who are pregnant, possibly pregnant, or lactating, or who plan to become pregnant
8. Subjects who received blood products, including albumins, within 7 days prior to the screening examination
9. Subjects who received any investigational drug other than OPC-41061 within 30 days prior to the screening examination
10. Subjects who previously participated in this or any other study of OPC-41061 and received OPC-41061
11. Subjects otherwise judged by the investigator or subinvestigator to be inappropriate for inclusion in the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2007-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Saito, Study Director — Division of New Product Evalution and Development
Locations (7):
- Japan (7):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyusyu Region
  - Tohoku Region

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo, 1 tablet a day
- OPC-41061 7.5 mg: 7.5 mg, 1 tablet a day
- OPC-41061 15 mg: 15 mg, 1 tablet a day
- OPC-41061 30 mg: 30 mg, 1 tablet a day
Period: Overall Study
Arm/Group | Placebo | OPC-41061 7.5 mg | OPC-41061 15 mg | OPC-41061 30 mg
Started | 27 | 26 | 25 | 26
Completed | 23 | 20 | 24 | 21
Not Completed | 4 | 6 | 1 | 5
Not completed — Adverse Event | 1 | 1 | 1 | 3
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 2
Not completed — Resolution of all hepatic edema findings | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 2 subjects (1 of placebo and 1 of OPC-41061 30 mg) were excluded by GCP deviation.
  1 subject (OPC-41061 7.5 mg) was excluded by receiving a dose 7 times higher than specified daily dose.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | OPC-41061 7.5 mg | OPC-41061 15 mg | OPC-41061 30 mg | Total
Number analyzed (Participants) | 26 | 25 | 25 | 25 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (10.1) | 64.5 (9.4) | 64.8 (9.7) | 62.8 (10.4) | 63.9 (9.8)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 11 | 11 | 13 | 48
  >=65 years | 13 | 14 | 14 | 12 | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 4 | 10 | 30
  Male | 17 | 18 | 21 | 15 | 71
Region of Enrollment [Number; unit: participants]
  Japan | 26 | 25 | 25 | 25 | 101

OUTCOME MEASURES:

1. Primary Outcome: Body Weight (Amount of Change)
Description: Changes in body wight from baseline at the final timepoint (LOCF). A linear regression model using changes in body weight from baseline at the final timepoint as the criterion variable and dose as the explanatory variable was fitted to the dataset.
Time Frame: Baseline, Day 7 or at the discontied of treatment
Population: Full Analysis Set; LOCF
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Placebo | OPC-41061 7.5 mg | OPC-41061 15 mg | OPC-41061 30 mg
Number analyzed (Participants) | 26 | 25 | 25 | 25
Kg | -0.68 (2.50) | -2.31 (2.35) | -1.88 (2.45) | -1.67 (1.46)
Statistical Analysis 1: Comparison: Placebo vs OPC-41061 7.5 mg vs OPC-41061 15 mg vs OPC-41061 30 mg; A linear regression model using change in body weight from baseline at the final timepoint as the criterion variable and dose as the explanatory variable was fitted to the dataset. The null hypothesis of whether the regression coefficient is zero (analysis using t-statistics) was tested at a two-tailed significance level of 0.05, and estimated values for the slope and 95% confidence interval were calculated; Test type: Superiority or Other; p = 0.3167, Regression, Linear; Slope = -0.021, 95% CI 2-sided [-0.061 to 0.020], Standard Error of Mean 0.020

2. Secondary Outcome: Abdominal Circumference
Description: Change in abdominal circumference from baseline (LOCF)
Time Frame: Baseline, Day 7 or at the discontied of treatment
Population: Full Analysis Set; LOCF
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo | OPC-41061 7.5 mg | OPC-41061 15 mg | OPC-41061 30 mg
Number analyzed (Participants) | 26 | 25 | 25 | 25
cm | -1.39 (3.16) | -2.98 (3.22) | -2.42 (3.96) | -2.62 (2.83)

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Placebo | OPC-41061 7.5 mg | OPC-41061 15 mg | OPC-41061 30 mg
Serious Adverse Events (participants affected / at risk) | 5/26 | 0/25 | 1/25 | 3/25
Other Adverse Events (participants affected / at risk) | 18/26 | 20/25 | 19/25 | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=26) | OPC-41061 7.5 mg (N=25) | OPC-41061 15 mg (N=25) | OPC-41061 30 mg (N=25)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic Failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hepatorenal Syndrome (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis B (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal Impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shock Haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=26) | OPC-41061 7.5 mg (N=25) | OPC-41061 15 mg (N=25) | OPC-41061 30 mg (N=25)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Supraventricular Extrasystoles (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 5 (7) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 5 (6) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (4)
Thirst (General disorders) | 1 (1) | 6 (6) | 14 (14) | 15 (15)
Malaise (General disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
Pyrexia (General disorders) | 3 (3) | 2 (2) | 3 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Blood Alkaline Phosphatase Increased (Investigations) | 1 (1) | 6 (6) | 3 (3) | 2 (2)
Blood Uric Acid Increased (Investigations) | 1 (1) | 3 (4) | 4 (4) | 5 (5)
Blood Bilirubin Increased (Investigations) | 5 (5) | 1 (1) | 1 (1) | 3 (3)
Blood Osmolarity Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Blood Urea Increased (Investigations) | 4 (4) | 4 (4) | 4 (4) | 3 (3)
Blood Creatinine Increased (Investigations) | 3 (3) | 2 (2) | 3 (3) | 2 (2)
Aspartate Aminotransferase Increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Blood Potassium Increased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Blood Pressure Decreased (Investigations) | 0 (0) | 2 (2) | 1 (3) | 1 (1)
Blood Sodium Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood Urine Present (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Platelet Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood Glucose Increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 6 (6) | 6 (6)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 8 (8) | 5 (5) | 12 (12)
Renal Impairment (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No